CLINICAL TRIAL: NCT00056355
Title: A Single Arm Study of Extracorporeal Photoimmune Therapy With Uvadex For Corticosteroid Sparing in Patients With Corticosteroid-Dependent Crohn's Disease Who May Also Be Refractory or Intolerant to Immunosuppressants and/or Anti-Tumor Necrosis Factor Agen
Brief Title: Extracorporeal Photopheresis to Maintain Symptoms Remission During Steroid Withdrawal in Patients With Steroid-Dependent Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030117; 03-I-0117
Record Dates: First submitted 2003-03-10; First posted 2003-03-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Crohn Disease
Keywords: Pheresis; Cytokine; Lymphocyte; Remission; Ultraviolet A Light; Crohn's Disease; Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Methoxsalen

INTERVENTIONS:
Drug: UVADEX and UVAR XTS Photopheresis System

SUMMARY:
This study will examine the safety and effectiveness of extracorporeal photopheresis (ECP) in controlling Crohn's disease symptoms as patients taper their corticosteroid dose. Crohn's disease is a chronic inflammatory bowel disease. Patients commonly have chronic diarrhea with abdominal pain, loss of appetite and weight loss. Acute disease flares are treated with large doses of corticosteroids, but long-term use of these drugs can have harmful side effects. ECP (described below), is approved to treat skin symptoms associated with a type of cancer called cutaneous T-cell lymphoma and has been used experimentally in conditions involving abnormal inflammation.

Patients 18 years of age and older who have had Crohn's disease for at least 6 months, who are corticosteroid-dependent, and whose symptoms are controlled well enough so that their Crohn's Disease Activity Index (CDAI) is less than 220, may be eligible for this study. Candidates will be screened with a medical history and review of medical records, physical examination, electrocardiogram, blood tests, urine pregnancy test for women of childbearing potential, and a questionnaire about how Crohn's disease affects their life and activities.

Patients with a CDAI score of less than 150 will begin ECP treatments as soon as possible. Those with scores from 150 to 219 will have their corticosteroid dose increased enough to bring their CDAI score to below 150 before beginning ECP. Patients who do not achieve a CDAI of less than 150 after 4 to 6 weeks of increased corticosteroids will be excluded from the study.

Participants will have ECP treatments for 2 consecutive days every 2 weeks for 24 weeks, for a total of 26 treatments. For ECP, patients undergo leukapheresis, a method of collecting large numbers of white blood cells, or leukocytes-cells that may be responsible for many of the medical problems in Crohn's disease. Whole blood is collected through a needle in an arm vein, similar to donating a unit of blood. The blood flows through a machine that separates it into its components by spinning. The white cells are removed and collected in a plastic bag, and the red blood cells and plasma are returned to the patient's bloodstream through the same needle. The collected white cells are mixed with a drug called UVADEX® (Registered Trademark), exposed to ultraviolet (UVA) light, and then returned to the patients' bloodstream. (The UVADEX allows the blood cells to absorb more UVA.) The UVA changes the cells in a way that, once they are back in the body, they cause changes in other cells like them. Each ECP treatment takes 3 to 4 hours. On the first day of each 2-day treatment, patients will undergo a review of symptoms, check of vital signs, and blood draw. They will complete a CDAI diary for 7 days before the first of the two ECP treatments and a questionnaire about their life and activities at 4-week intervals. During the ECP treatment period, corticosteroids will be slowly reduced as long as disease symptoms do not worsen.

Patients whose disease remains under control with cessation of all steroids may begin maintenance ECP, 2 days in a row every 4 weeks for an additional 20 weeks (another 10 treatments), with the same follow-up as described above, and a full physical examination 4 weeks after the final treatment. Patients who were able to reduce, but not stop, steroid treatment may be considered for maintenance therapy if it is thought that continuing treatment may enable further reduction of steroids. Patients whose disease symptoms worsen with ECP or who have not been able to decrease their steroid dose will not be eligible for maintenance therapy and their participation in the study will end.

DETAILED DESCRIPTION:
This protocol aims to measure the safety and effectiveness of extracorporeal photopheresis (ECP) therapy for maintaining remission of symptoms during withdrawal of corticosteroids from patients with steroid-dependent Crohn's disease. Potential subjects will be asymptomatic or have a low level of symptoms that respond to an increase in their steroid dose; furthermore potential subjects will be dependent on steroids to control their symptoms and have a history of failing other immunosuppressive drugs to control their symptoms.

This is an unblinded, single-arm study of ECP in Crohn's disease. This trial will use ECP twice a week every two weeks over 24 weeks during which time the dose of corticosteroids will be tapered. If the corticosteroids are able to be withdrawn without an increase in symptoms, then subjects may be eligible for further ECP (twice a week every four weeks over 24 weeks) as a maintenance regimen.

Outcome parameters include the rates of complete and partial steroid tapering while maintaining remission, the rates of adverse events, and secondary clinical outcomes such as duration of response, rate of and time to relapse, and changes in symptom index scores. In addition, the NIH will perform a substudy that includes serial colonoscopy to measure cytokine and cell population changes in mononuclear cells extracted from biopsies.

The long-term goals of this study are to test the safety and efficacy of ECP as a steroid-sparing and remittive therapy in Crohn's disease, to determine the immune response it effects in the gut mucosa, and identify factors associated with responders versus non-responders to ECP.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet each of the following criteria to be eligible for enrollment in this study.

1. Patients with Crohn's disease of at least 6 months duration (with colitis, ileitis, or ileocolitis) confirmed by radiography or endoscopy.
2. Patient must have a CDAI score less than 220.
3. Patients with corticosteroid-dependent Crohn's disease who have failed at least one attempt at corticosteroid tapering within the previous 6 months. Corticosteroid-dependent patients are defined as those patients who have relapse of Crohn's disease within 60 days following completion of corticosteroid treatment; OR during corticosteroid tapering at doses greater than or equal to 10 mg/day (prednisone equivalent); OR within 3 months following corticosteroid tapering, while receiving a corticosteroid dose greater than or equal to 10 mg/day.
4. Patients with a CDAI score of less than 150 MUST:

   * be on oral corticosteroids (other than oral budesonide) greater than or equal to 10 mg/day to be on oral corticosteroids (prednisone equivalent) for Crohn's disease;
   * be on a stable dose of oral corticosteroids (other than oral budesonide) for at least 2 weeks prior to screening;
   * have had clinically inactive Crohn's disease for at least 2 weeks prior to screening.

   OR

   Patients with a CDAI score of greater than or equal to 150 to less than 220 MUST:
   * be on oral corticosteroids (othern than oral budesonide) greater than or equal to 10 mg/day to less than or equal to 40 mg/day (prednisone equivalent) for Crohn's disease;
   * have had no worse than mild disease for at least 2 weeks prior to screening.
5. Patients on aminosalicylates must have been on a stable dose for at least 4 weeks prior to screening; and patients on the immunosuppressants, azathioprine, 6-mercaptopurine, or methotrexate must have been on a stable dose for at least 8 weeks prior to screening.
6. Patients not using aminosalicylates must have discontinued treatment at least 4 weeks prior to screening. Patients not using immunosuppressants such as azathioprine, 6-mercaptopurine, or methotrexate must have discontinued treatment at least 4 weeks prior to screening. Patients who had been receiving infliximab must have stopped therapy at least 8 weeks prior to screening. Patients who had been receiving adalimumab, cyclosporine, tacrolimus, or mycophenolate mofetil must have stopped therapy for at least 4 weeks prior to screening.
7. Patients who have incidental (e.g. perianal) fistulae are permitted, provided:

   * patients have predominantly luminal Crohn's disease, and
   * fistulae are not associated with retention.
8. Patient's platelet count must be greater than or equal to 20,000/cmm.
9. Female patients must be one of the following: postmenopausal, surgically incapable of bearing children, practicing an acceptable method of birth control (acceptable methods may include hormonal contraceptives, intrauterine device, and spermicide and barrier). Abstinence or partner/spouse sterility may also qualify at the Investigator's discretion. If a female patient is of childbearing potential she must have a negative urine pregnancy test at screening.
10. Patients must be able and willing to comply with all study procedures.
11. Signed informed consent must be obtained prior to conducting any study procedures.
12. Patients must be men and women greater than or equal to 18 years of age.
13. Patients must have a body weight greater than or equal to 40 kg (88 lb).

EXCLUSION CRITERIA:

The presence of any of the following criteria will exclude the patient from from participating in the study:

1. Patients with symptomatic intestinal strictures.
2. Patients with local manifestations of Crohn's disease such as abscesses, or disease manifestations for which surgery might be indicated, or which might preclude utilization of a CDAI to assess response to therapy (such as "short gut" syndrome).
3. Patients with stomas.
4. Patients with rectovaginal fistulae.
5. Patients who require antibiotics for the treatment of Crohn's disease.
6. Patients using oral budesonide.
7. Patients with diarrhea, due to conditions other than inflammatory Crohn's disease (e.g. bacterial or parasitic gastroenteritis, bile salt diarrhea, or bacterial overgrowth).
8. Patients who are concomitantly using an anti-TNF agent, antibiotics, nonsteroidal anti-inflammatory drugs (NSAIDs), cyclosporine, tacrolimus, mycophenolate mofetil, or investigational therapies.
9. Patients unable to tolerate the extracorporeal volume shifts associated with ECP treatment due to the presence of any of the following conditions: uncompensated congestive heart failure, pulmonary edema, severe chronic obstructive pulmonary disease, severe asthma, renal failure, or hepatic failure.
10. Patients with a poor tolerability of venipuncture or a lack of adequate venous access for required blood sampling.
11. Patients receiving total parenteral nutrition (TPN), as the sole source of nutrition, within 3 weeks of screening.
12. Patients with hypersensitivity or allergy to psoralen (methoxsalen).
13. Patients with hypersensitivity or allergy to both heparin and citrate products.
14. Patients with active bleeding.
15. Females who are pregnant and/or lactating.
16. Patients must not have been enrolled in any investigational study for 30 days prior to enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2003-03; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Edelson R, Berger C, Gasparro F, Jegasothy B, Heald P, Wintroub B, Vonderheid E, Knobler R, Wolff K, Plewig G, et al. Treatment of cutaneous T-cell lymphoma by extracorporeal photochemotherapy. Preliminary results. N Engl J Med. 1987 Feb 5;316(6):297-303. doi: 10.1056/NEJM198702053160603. PMID 3543674
- [Background] Schafer-Korting M, Korting HC. Intraindividual variations of 8-methoxypsoralen plasma levels. Arch Dermatol Res. 1982;272(1-2):1-7. doi: 10.1007/BF00510387. PMID 7165313
- [Background] Herfst MJ, De Wolff FA. Intraindividual and interindividual variability in 8-methoxypsoralen kinetics and effect in psoriatic patients. Clin Pharmacol Ther. 1983 Jul;34(1):117-24. doi: 10.1038/clpt.1983.139. PMID 6861433